CLINICAL TRIAL: NCT07233122
Title: MRI Vs Conventional Radiography in Assessing Knee Hemophilic Arthropathy : A Scoring Based Approach
Brief Title: MRI Role in Knee Hemophilic Arthopathy
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, kerolos wagdy maurice morid, Principal Investigator, Assiut University
Other Study IDs: MRI in Hemophilic Arthopathy
Record Dates: First submitted 2025-09-19; First posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: MRI; Hemophilia; Arthropathy Hemophilic; Arthropathy of Knee
MeSH Terms: conditions — Hemophilia A

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MRI in Knee Hemophilic Arthopathy: Participants diagnosed with hemophilia and clinical suspicion of knee arthropathy will undergo magnetic resonance imaging (MRI) of the affected knee. MRI will be performed using standardized sequences to evaluate joint changes, including synovial hypertrophy, hemosiderin deposition, cartilage thinning, and bone damage. Findings will be scored using the International Prophylaxis Study Group (IPSG) MRI scoring system.
- Xray in Knee Hemophilic Arthropathy: Participants diagnosed with hemophilia and clinical suspicion of knee arthropathy will undergo conventional radiography (X-ray) of the affected knee. Standard anteroposterior and lateral views will be obtained to evaluate joint changes, including joint space narrowing, osteoporosis, subchondral cysts, erosions, and bone deformities. Findings will be scored using the Pettersson X-ray scoring system.

SUMMARY:
The aim of this study is to assess role of MRI in detecting synovial, cartilaginous , osseous abnormalities ، bleeding inside knee joint and to use a system for assessing HA as support for therapeutic regimes and for monitoring response to therapy .

DETAILED DESCRIPTION:
Hemophilia is a mostly inherited genetic disorder caused by a complete or partial deficiency of coagulation factors VIII or IX, which impairs the body's ability to form blood clots-a process necessary to stop bleeding. This results in prolonged bleeding after injury, easy bruising, and an increased risk of internal bleeding, particularly within joints or the brain.

Hemophilic arthropathy (HA), caused by recurrent hemarthrosis, is the most common musculoskeletal manifestation of hemophilia and one of the most disabling complications of the disease. It can lead to severe pain, deformity, destruction of the joint, debilitating arthritis, and permanent joint damage.

Clinical assessment plays only a minor role in detecting the early stages of HA, as early clinical signs are often nonspecific and of limited value in quantifying disease involvement. Conventional radiographs mainly detect bone lesions that appear in advanced HA, but they cannot identify early changes such as synovial hypertrophy or focal cartilage destruction. Computed tomography (CT) is highly sensitive for detecting bone changes, but it provides limited information on soft tissue involvement and requires a relatively high dose of ionizing radiation.

By contrast, magnetic resonance imaging (MRI) offers superior soft tissue contrast, allowing detailed evaluation of hemophilic joints and visualization of synovial and cartilaginous abnormalities.

T1-weighted imaging: evaluates bone marrow, joint anatomy, and subchondral changes.

T2 fat-suppressed imaging: useful for detecting synovitis and joint effusion.

Gradient echo (GRE) or susceptibility-weighted imaging (SWI): detect chronic blood products (hemosiderin), with SWI being more sensitive and able to identify earlier blood deposits.

Several scoring systems exist for the assessment of hemophilic arthropathy, including the European scoring system and the International Prophylaxis Study Group (IPSG) MRI scale. The IPSG system provides more detailed scoring and greater sensitivity for early disease, including subtle synovial changes. For radiographs, the most widely used system is the Pettersson radiographic scoring system.

In this study, the investigators will use the IPSG MRI scoring system and the Pettersson X-ray scoring system to evaluate hemophilic arthropathy, with the aim of improving grading, management, and follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient ( more than 18 years old ) diagnosed as Haemophilia with history of bleeding in knee joint more than once

Exclusion Criteria:

* *contraindications for MRI such as claustrophobia , metallic foriegn body carriers , cardiac pacemaker

  * patient refused the exam
  * Pregnant female patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include patients diagnosed with hemophilia A or hemophilia B who are at risk of, or clinically suspected to have, hemophilic arthropathy of the knee joint. Participants will be recruited from hematology and orthopedic clinics.
  Eligible participants will undergo knee MRI to assess for:
  Synovial abnormalities (e.g., hypertrophy, hemosiderin deposition)
  Cartilaginous changes (thinning, erosions)
  Osseous changes (subchondral cysts, bone erosions, marrow changes)
  Intra-articular bleeding
  MRI scoring systems will be applied to quantify disease severity and to evaluate the role of MRI as a tool for supporting therapeutic decisions and monitoring treatment response.
Sampling Method: Non-Probability Sample
Enrollment: 95 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
International Prophylaxis Study Group (IPSG) MRI Score for Hemophilic Arthropathy | After completion of MRI scanning session (within the same study visit). Overall Study Duration: 2 years (for recruitment, imaging, and data analysis).
  Assessment of knee hemophilic arthropathy severity using the International Prophylaxis Study Group (IPSG) MRI scoring system. This scoring system evaluates early and advanced joint changes such as synovial hypertrophy, hemosiderin deposition, and cartilage/bone damage.

SECONDARY OUTCOMES:
Pettersson X-ray Score for Hemophilic Arthropathy | After completion of X-ray scanning session (within the same study visit). Overall Study Duration: 2 years (including recruitment, imaging, and data analysis).
  Assessment of knee hemophilic arthropathy severity using the Pettersson X-ray scoring system. This system evaluates joint space narrowing, osteoporosis, subchondral cysts, erosions, and bone deformities to quantify the degree of arthropathy.
Agreement Between MRI and X-ray Scoring Systems in Hemophilic Arthropathy | After completion of MRI and X-ray scanning sessions (within the same study visit). Overall study duration: 2 years (including recruitment, imaging, and data analysis).
  To evaluate the agreement between the International Prophylaxis Study Group (IPSG) MRI score and the Pettersson X-ray score in assessing the severity of knee hemophilic arthropathy. This outcome will determine the level of concordance between the two imaging modalities in detecting joint changes.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Ibad HA, de Cesar Netto C, Shakoor D, Sisniega A, Liu SZ, Siewerdsen JH, Carrino JA, Zbijewski W, Demehri S. Computed Tomography: State-of-the-Art Advancements in Musculoskeletal Imaging. Invest Radiol. 2023 Jan 1;58(1):99-110. doi: 10.1097/RLI.0000000000000908. Epub 2022 Aug 16. PMID 35976763
- [Result] Foppen W, van der Schaaf IC, Beek FJA, Mali WPTM, Fischer K. MRI predicts 5-year joint bleeding and development of arthropathy on radiographs in hemophilia. Blood Adv. 2020 Jan 14;4(1):113-121. doi: 10.1182/bloodadvances.2019001238. PMID 31917842
- [Result] Lundin B, Manco-Johnson ML, Ignas DM, Moineddin R, Blanchette VS, Dunn AL, Gibikote SV, Keshava SN, Ljung R, Manco-Johnson MJ, Miller SF, Rivard GE, Doria AS; International Prophylaxis Study Group. An MRI scale for assessment of haemophilic arthropathy from the International Prophylaxis Study Group. Haemophilia. 2012 Nov;18(6):962-70. doi: 10.1111/j.1365-2516.2012.02883.x. Epub 2012 Jul 5. PMID 22765835
- [Result] Haacke EM, Mittal S, Wu Z, Neelavalli J, Cheng YC. Susceptibility-weighted imaging: technical aspects and clinical applications, part 1. AJNR Am J Neuroradiol. 2009 Jan;30(1):19-30. doi: 10.3174/ajnr.A1400. Epub 2008 Nov 27. PMID 19039041
- [Result] Kim HK, Zbojniewicz AM, Merrow AC, Cheon JE, Kim IO, Emery KH. MR findings of synovial disease in children and young adults: Part 1. Pediatr Radiol. 2011 Apr;41(4):495-511; quiz 545-6. doi: 10.1007/s00247-011-1971-0. Epub 2011 Feb 22. PMID 21337125